CLINICAL TRIAL: NCT01392157
Title: Acceptability and Continuation Rate of Implanon in a Brazilian Public Sector
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Luis Bahamondes, MD Medical Doctor, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/2011/PC
Record Dates: First submitted 2011-06-16; First posted 2011-07-12 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Contraceptive Usage; Bleeding Due to Intrauterine Contraceptive Device
MeSH Terms: conditions — Contraception Behavior | interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- copper intrauterine device (Active Comparator): 100 women will be allocated to receive a TCu380A intrauterine device
  Interventions: Device: copper-releasing intrauterine device; Device: ENG-releasing implant; Device: LNG-releasing intrauterine system; Device: LNG-IUS
- LNG-releasing intrauterine system (Active Comparator): 100 women were allocated to receive a LNG-IUS
  Interventions: Device: ENG-releasing implant; Device: LNG-releasing intrauterine system; Device: LNG-IUS
- ENG-releasing implant (Active Comparator): 100 women will receive an LNG-IUS
  Interventions: Device: ENG-releasing implant; Device: LNG-releasing intrauterine system; Device: LNG-IUS

INTERVENTIONS:
Device: copper-releasing intrauterine device — 100 women received a 380 mm2 of copper releasing intrauterine device
  Other Names: Optima, Injeflex, Brazil
  Arms: copper intrauterine device
Device: ENG-releasing implant — 60 mcg/day releasing etonogestrel implant
  Other Names: Implanion, MSD, Os, The Nedherland
Device: LNG-releasing intrauterine system — a LNG-IUS releasing 20 mcd/day of LNG
  Other Names: Mirena, Bayer Oy, Turku, Finland
Device: LNG-IUS — 100 women will receive an LNG-IUS
  Other Names: Mirena, Bayer Oy, Turku, Finland

SUMMARY:
The main side-effect of Implanon is the changes induces in bleeding patterns including amenorrhea, infrequent to irregular bleeding and frequent and prolonged bleeding; without any previous symptom and it was characterized as "breakthrough bleeding" (BTB). BTB is the main causes of early discontinuations. Unfortunately, there is no indication to predict prior to insertion what sort of bleeding pattern any individual woman may have after insertion and the proposed treatments were disappointed. Nevertheless, previous studies with other progestin-only contraceptives (including Implanon) provide evidence that the provision of adequate and intensive counseling to potential users and new acceptors about bleeding changes can help to improve method continuation.

The availability of Implanon in the public sector could help in the development of strategies to introduce the method in the public sector network and the training of medical residents.

DETAILED DESCRIPTION:
100 women were either allocated to received Implanon contraceptive implant, the LNG-IUS or TCu380A copper-IUD. The women were allocated according to their preference on each of the contraceptive methods.

half of the women will receive the common counseling at the clinic and the other 50% will receive intense counselling about menstrual changes induced by these three contraceptive methods. The continuation rate up to one year will be evaluated through life-table analysis

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 40 years
* New users of Implanon, IUDs and the LNG-IUS TCu380A

Exclusion Criteria:

* Contraindications to contraceptive methods

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Assessment of acceptability of Implanon in comparison to the TCu380A IUD and the LNG-IUS | Participants will receive counseling before admission and at 12 months after
  All the acceptors (contraceptive implants, the LNG-IUS and the copper IUD) will be follow for up to one year and we will record all the adverse events and mainly all the discontinuations due to bleeding irregularities, to compare one group to other and the half of the women who will receive intense counseling in comparison to the women with regular counseling at the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Bahamondes, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Modesto W, Bahamondes MV, Bahamondes L. A randomized clinical trial of the effect of intensive versus non-intensive counselling on discontinuation rates due to bleeding disturbances of three long-acting reversible contraceptives. Hum Reprod. 2014 Jul;29(7):1393-9. doi: 10.1093/humrep/deu089. Epub 2014 May 8. PMID 24812309